CLINICAL TRIAL: NCT03393169
Title: Evaluation of Post-operative Morbidity and Mortality After Cardiac Surgery Performed in Bichat Hospital
Brief Title: Postoperative Morbidity and Mortality After Cardiac Surgery
Acronym: Cardiobase
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: Cardiobase
Record Dates: First submitted 2017-05-02; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2017-12

CONDITIONS: Cardiac Surgery Under Extra Corporeal Circulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The local database results from a joint initiative of anesthesic, cardiology and cardiac surgery departements.Its purpose is to record in an exhaustive fashion all the interventions of cardiac surgery performed under extracorporeal circulation in adults at Bichat hospital.This database includes the preoperative characteristics of the patients, the type of surgery, the post-operative complications and the in-hospital mortality. The purpose of this observational study is to evaluate in-hospital morbidity and mortality for all types of cardiac surgery interventions and to analyze it according to the characteristics of the patients and the type of intervention.

DETAILED DESCRIPTION:
The operative mortality is a key point of the risk-to-benefit ratio analysis before considering cardiac surgery. Operative risk evaluation in a single surgical center is a part of medical care quality assessment. It must be interpreted in the light of the local specificities, in particular the characteristics of the patients and the types of surgery. The local database results from a joint initiative of anesthesic, cardiology and cardiac surgery departements.Its purpose is to record in an exhaustive fashion all the interventions of cardiac surgery performed under extracorporeal circulation in adults at Bichat hospital.This database includes the preoperative characteristics of the patients, the type of surgery, the post-operative complications and the in-hospital mortality. The purpose of this observational study is to evaluate in-hospital morbidity and mortality according to the characteristics of the patients and the type of intervention. study population : inclusion criteria : patient 18 years or older with legal capacity, patients with non-objection to record his/her medical data during hospitalization. Methods: this is an observational prospective and monocentric study. The main objective is to report in-hospital mortality for all types of cardiac surgery performed in Bichat hospital . The secondary objectives are :1) to collect post-operative complications such as hemorrhagic or thromboembolic events or surgery site infections; 2) to analyze mortality rate and post-operative morbidities according to the type of surgery and the main patients' characteristics . 3) to calculate validated and currents risk score such as EuroSCORE I and II for each patient.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older and has legal capacity - cardiac surgery under extra corporeal circulation
* non objection to record medical information during hospitalization

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients , 18 years old and older, with a cardiac surgery under extra corporeal circulation in Bichat Hospital
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2006-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days
  All-cause mortality is assessed during in-hospital stay and 30 days after the date of surgery

SECONDARY OUTCOMES:
Postoperative organ failure | 30 days
  Cardiac with inotropic or mechanical support, renal failure or need for dialysis, pulmonary (mechanical ventilation duration), neurologic or digestive complications
Bleeding complications | 30 days
  Total blood loss, transfusion requirements, surgical reexploration
Arrhythmias | 30 days
  Atrial fibrillation, ventricular tachycardia
Conductions disturbances | 30 days
  Need for pace maker implantation
Myocardial injury | 30 days
  Troponin I release (ng/mL)
Postoperative sepsis | 30 days
  Pneumonia, septicemia and endocarditis, surgical site infection
Risk score calculation: Euroscore II | 30 days
  Calculation with all the items required by the published and validated equation
Length of stay | 30 days
  Length of stay in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Bernard IUNG, MD., Study Director — Assistance Publique Hopitaux de Paris
Locations (1):
- département de cardiologie et d'anesthésie réanimation Hôpital Bichat 46 rue Henri Huchard, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
with others French University Hospitals (Rennes, Nantes, Paris (PITIE SALPETRIERE) , Bordeaux)